CLINICAL TRIAL: NCT02605343
Title: Prospective Observational Clinical Study to Evaluate Patient Outcomes Following Pharmacogenetic Testing of Patients Undergoing Elective Surgical Procedures Compared to Historical Data
Brief Title: Prospective Observational Clinical Study to Evaluate Patient Outcomes Following Pharmacogenetic Testing of Patients Undergoing Elective Surgical Procedures
Status: Completed | Type: Observational
Sponsor: AltheaDx (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CLP0006
Record Dates: First submitted 2015-11-06; First posted 2015-11-16 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2015-11

CONDITIONS: Acute Pain; Surgery
Keywords: PGx; pharmacogenetic testing; Pain Management; AltheaDx; Post-Operative Pain Management
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NeuroIDgenetix-guided Pain Management: The medical provider for the NeuroIDgenetix-guided group will make post-operative pain management recommendations based on test results. Patient outcomes, narcotic consumption, opioid-related adverse effects, time to mobilization, number of adverse drug events and number of hospital and/or medical visits will be measured throughout the study.
  Interventions: Other: NeuroIDgenetix Test Panel
- Historical Control: The retrospective chart review will utilize patient outcomes from patients meeting the study inclusion/exclusion criteria. The medical provider for the control group will not have received the NeuroIDgenetix Test Panel results and would have made post-operative pain management recommendations per standard of care.

INTERVENTIONS:
Other: NeuroIDgenetix Test Panel — The NeuroIDgenetix Test Panel is used to make recommendations on post-operative pain medication therapy that may be impacted by the genetic background of the patient.
  Other Names: IDgenetix Neuro Test; PGx Testing
  Groups: NeuroIDgenetix-guided Pain Management

SUMMARY:
The purpose of this study is to evaluate the effect of pharmacogenetics (PGx) guided treatment when implemented into the pre-operative process for patients undergoing bowel surgery, major urologic procedure, or major ventral hernia repair and requiring post-operative acute pain management in an inpatient basis, as compared to a group of subjects with the same attributes without the guidance of PGx testing (historical control group). This study will also evaluate the frequency with which the standard analgesic care plan is adjusted by test results.

DETAILED DESCRIPTION:
The incidence of opioid-related adverse drug events can reach as high as 50% in surgical patients and poor pain management is a significant risk factor for early readmission. In addition, the rate of non- response to certain analgesics is double in patients who are poor metabolizers as demonstrated by mutations in both CPY26D alleles. There is a growing body of literature that indicate that ineffective acute pain management contributes significantly to the risk of chronic pain syndromes. Genetics and drug interactions can alter both the pharmacokinetics and pharmacodynamics of a multitude of drug compounds and in turn influence both the safety and efficacy of selected therapeutic regimens.

Pharmacogenetic-guided therapy selection can enhance patient response by facilitating the selection of the most appropriate medication at the most effective dose in the shortest possible time.

In this prospective, observational, single-blind study, the investigators will evaluate the clinical impact of pharmacogenetics-guided treatment on patient well-being as determined by post-op pain assessments and the frequency of changes in analgesics predicted by testing results. Additionally, the impact of PGx-guided treatment on narcotic consumption, time to mobilization, number of adverse events, length of stay, and re-admission rates compared to historical data will be evaluated during the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over the age of 18
* Presenting to the site for a prep-op visit prior to undergoing a major bowel surgery, major urologic procedure or major ventral hernia repair. The pre-op visit must occur at least 3 days prior to the surgical procedure.
* Willing and able to comply with study procedures
* Able to provide written informed consent

Exclusion Criteria:

* Unwilling or unable to provide written informed consent and to comply with study procedures;
* Unwilling or unable to provide buccal swab sample
* History of chronic renal dysfunction, Chronic Kidney Disease (Stage 4 or 5);
* New York Heart Classification >3
* Abnormal hepatic function within the last 2 years (INR >1.2 not attributable to anticoagulant medications, AST/aspartate aminotransferase or ALT/alanine aminotransferase >1.5x normal, or suspected cirrhosis);
* History of malabsorption (short gut syndrome);
* Gastric or small bowel surgery less than 3 months prior to study enrollment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the site for a prep-op visit prior to undergoing a major bowel surgery, major urologic procedure or major ventral hernia repair. The pre-op visit must occur at least 3 days prior to the surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comparison of patient well-being measured by OBAS score between the two study groups. | From date of surgery until last follow-up visit, assessed at 30 days post-surgery
  Comparison of patient well-being between experimental and control group as measured by Overall Benefit of Analgesics (OBAS) score.
Comparison of length of post-surgical hospital stay between the two study groups | From date of surgery until hospital discharge, assessed up to 1 month
  Comparison of duration of post-surgical hospital stay between experimental and control group.
Comparison of patient well-being measured by BPI score between the two study groups | From date of surgery until last follow-up visit, assessed at 30 days post-surgery
  Comparison of patient well-being between experimental and control group as measured by Brief Pain Inventory-Short Form score.

SECONDARY OUTCOMES:
Comparison of post-operative narcotic consumption between the two study groups | From date of surgery until last follow-up visit, assessed at 30 days post-surgery
  Comparison of post-operative narcotic consumption between the two study groups
Comparison of time to mobilization between the two study groups | From date of surgery to mobilization, assessed up to 30 days post-surgery
  Comparison of time to mobilization between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Senagore, MD, Principal Investigator — University Hospitals Case Medical Centers
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No